CLINICAL TRIAL: NCT06496841
Title: A Comparison of Transnasal Versus Ultrasound-guided Suprazygomatic Approaches for Sphenopalatine Ganglion Blocks in Persistent Idiopathic Facial Pain
Brief Title: Transnasal Versus Suprazygomatic SPG Block in Persistant Idiopathic Facial Pain
Status: Completed | Type: Observational
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, Principal investigator, Diskapi Teaching and Research Hospital
Other Study IDs: SPG block
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Headache; Persistent Idiopathic Facial Pain
Keywords: headache; ultrasonography; sphenopalatine ganglion block; Persistent Idiopathic Facial Pain
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transnasal sphenopalatine ganglion block group: transnasal administration of lidocaine to the sphenopalatine ganglion
  Interventions: Drug: Transnasal Sphenopalatine ganglion block
- Ultrasound-guided suprazygomatic sphenopalatine ganglion block group: ultrasound-guided suprazygomatic approach
  Interventions: Drug: Ultrasound-guided suprazygomatic sphenopalatine ganglion block

INTERVENTIONS:
Drug: Transnasal Sphenopalatine ganglion block — The transnasal approach to the sphenopalatine ganglion block allows for non-invasive access to the sphenopalatine ganglion, which is located deep in the nasopharynx in a recess posterior to the middle turbinate. A long cotton swab is inserted posterior to the nasopharynx until it is properly seated, and 2 mL of 2% lidocaine is injected through the outer end of the swab and left for 30 minutes. Patients are monitored for any potential complications or adverse effects throughout the procedure and for a period of time afterwards.
  Groups: Transnasal sphenopalatine ganglion block group
Drug: Ultrasound-guided suprazygomatic sphenopalatine ganglion block — The ultrasound transducer is placed in the infrazygomatic area, above the maxilla, at approximately a 45 cephalad angle. With this transducer position, the ptrigopalatine fossa, bounded anteriorly by the maxilla and posteriorly by the pterygoid process, is visualized. A 25 gauge spinal needle is inserted 1 to 1.5 cm above the zygomatic arch and posterior to the posterior orbital rim and advanced through an out-of-plane approach to reach the pterigolapalatine fossa. After the aspiration test, 3 mL of 2% lidocaine is injected and the spread of the drug is monitored by ultrasound. Patients are monitored for possible side effects and complications.
  Groups: Ultrasound-guided suprazygomatic sphenopalatine ganglion block group

SUMMARY:
The International Headache Society defines persistent idiopathic facial pain (PIFP) as persistent facial pain that does not have the characteristics of cranial neuralgia, is blunt, persistent, persistent, bothersome and not attributable to another disorder. The management of persistent idiopathic facial pain (PIFP) is complex. The sphenopalatine ganglion (SPG) has been the target of interventional treatment of many facial pain syndromes. The sphenopalatine ganglion can be accessed by transnasal access and ultrasound or scopy guidance. In this study, datas compared the efficacy of transnasal approach and ultrasound-guided suprazigomatic approach in sphenopalatine ganglion block in patients with persistent idiopathic facial pain.

DETAILED DESCRIPTION:
Patients with chronic head and facial pain are frequently referred to us and some of these patients are persistent idiopathic facial pain patients who do not respond to conservative treatment. Various interventional treatment modalities can be applied to these patients. One of the treatments we frequently apply is sphenopalatine ganglion (SPG) blockage, which has an important place in the pathogenesis of chronic headache. The SPG is the target area for the treatment of cluster headache, migraine, postherpetic neuralgia, trigeminal neuralgia and other atypical facial pain syndromes due to its anatomical localisation and its role in the trigemino-cervical reflex. Although there are various techniques for SPG block, the simplest and most easily applicable is the transnasal approach and the traditional method is to apply a block with a cotton-tipped swab. Various local anaesthetics can be used, the most commonly used local anaesthetic is 2-3 ml of 2% or 10% lidocaine, usually administered through one nostril for 30 minutes. It is also possible to access SPG via the suprazygomatic route, and studies have shown that SPG block applied via the suprazygomatic route provides effective treatment of chronic headaches. In ultrasound-guided SPG block, after visualising the pterygopalatine fossa with USG, 3-4 mL of 2% lidocaine is administered to the area and blockage is achieved.

Our study was designed retrospectively. The primary aim of the study was to compare the efficacy of transnasal and suprazigomatic routes based on Numerical Rating Scale (NRS) pain scores by reviewing the files of patients who underwent sphenopalatine ganglion block for persistent idiopathic facial pain. The pain scores recorded before the procedure and one and four weeks after the procedure will be compared.

In this study, primary aim is to evaluate the efficacy of these two treatment modalities, with retrospectively evaluate the Visual Analogue Scale (VAS) score, HIT-6 (Headache Impact Test-6) score and headache diary data of the patients who have previously undergone these treatments in the pain clinic.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of persistent idiopathic facial pain according to ICHD-3 beta criteria
* Moderate to severe pain (pain of 6 or more on a numeric pain scale of 0-10)
* Persistence of pain for more than 6 months
* Pain unresponsive to conservative methods

Exclusion Criteria:

* Presence of secondary headache (tumor, bleeding, stroke, etc.)
* Cognitive impairment
* Hepatic or renal insufficiency
* Local or systemic infection
* Coagulopathy
* Patient refusal to accept treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients who underwent transnasal or ultrasound-guided suprazygomatic sphenopalatin ganglion block for persistant idiopathic facial pain
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-02 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | Change from baseline to 1st hour, 1st week and 4th weeks after treatment
  NRS is a pain screening Scale, in time using a 0-10 Scale, with zero meaning ''no pain'' and 10 meaning ''the worst pain imaginable''.

SECONDARY OUTCOMES:
HIT-6 (Headache impact test) | Change from baseline to 1st hour, 1st week and 4th weeks after treatment
  HIT-6 is a self-report questionnare designed to evaluate the impact of headache on quality of life. 49 or less: little or no impact, 50-55: some impact, 56-59. substantial impact, 60-78: severe impact

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Taylan Akkaya, MD, Study Director — Diskapi Teaching and Research Hospital; Ezgi Can, MD, Principal Investigator — Diskapi Teaching and Research Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided